CLINICAL TRIAL: NCT07001345
Title: Alveolar Ridge Preservation (ARP) Versus Spontaneous Healing in Large Buccal Bone Defects After Tooth Extraction in the Posterior Mandible
Brief Title: Alveolar Ridge Preservation Versus Spontaneous Healing
Acronym: ARP versus SH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Justin Pijpe, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL-009366
Record Dates: First submitted 2025-05-01; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Dental Implants, Single-tooth; Alveolar Ridge Preservation; Guided Bone Regeneration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARP with xenograft (Experimental): ARP with xenograft (Cerabone ® plus, Botiss Biomaterials GmbH, Zossen, Germany) covered by a native collagen membrane (Jason ® membrane, Botiss Biomaterials GmbH, Zossen, Germany) and delayed implant placement (4-6 months after extraction).
  Interventions: Procedure: Alveolar Ridge Reconstruction
- ARP with allograft (Experimental): ARP with a freeze dried bone allograft (Maxgraft®, Botiss Biomaterials GmbH, Zossen, Germany) covered by a native collagen membrane (Jason ® membrane, Botiss Biomaterials GmbH, Zossen, Germany) and delayed implant placement (4-6 months after extraction).
  Interventions: Procedure: Alveolar Ridge Reconstruction
- Spontaneous healing (No Intervention): spontaneous healing and delayed implant placement (4-6 months after tooth extraction).

INTERVENTIONS:
Procedure: Alveolar Ridge Reconstruction — Alveolar ridge preservation with either xenograft of allograft material
  Arms: ARP with allograft; ARP with xenograft

SUMMARY:
Rationale: To determine the effect of alveolar ridge preservation (ARP) versus spontaneous healing (SH) in large buccal bone defects in the posterior mandible.

Objective: To evaluate whether ARP using a xenograft (XG) (Cerabone plus) or an allograft (AG) (Maxgraft granules) covered by a membrane (Jason membrane) reduces the need for additional bone augmentation either prior to or during implant placement in the posterior mandible compared to spontaneous healing Study design: Prospective randomized clinical study with 10-year follow-up.

Study population:

Inclusion criteria: patients are 18 years or older and in need for extraction of a (pre)molar in the posterior mandible with at least one adjacent tooth and a buccal bone defect of >50%.

Exclusion criteria: the presence of active periodontal disease, uncontrolled diabetes mellitus, a history of or current use of chemotherapy or radiation in the head and neck area, history of or current use of medication related to osteonecrosis of the jaw, smoking (> 5 cigarettes a day, disability (physical and/or mental), making the patient unable to maintain basic oral health or follow the study protocol, pregnancy (in case of pregnancy, the treatment is postponed until after the delivery).

Intervention (if applicable): Atraumatic extraction of a (pre)molar in the posterior mandible will be performed. Patients will then be included based on the dimensions of the buccal bone defect (buccal bone defect of >50%). 66 patients will be randomly divided in either the XG group, the AG group or the SH group (control). In the ARP groups (XG and AG), following tooth extraction, ARP will be performed using either a XG (Cerabone plus) or an AG (Maxgraft granules), both covered by a membrane (Jason membrane). In the control group, the alveolus will be left for spontaneous healing, following tooth extraction. After 4-6 months, a cone bean computed tomography (CBCT) scan will be performed to determine the possibility of implant placement with or without additional augmentation. Implant placement will be performed in all groups with or without guided bone regeneration (GBR).

Main study parameters/endpoints: Frequency of additional augmentation at implant placement.

DETAILED DESCRIPTION:
Extraction of the teeth in the posterior region of the mandible may be an indication for the placement of dental implants. However, after extraction of the teeth, the alveolar ridge undergoes changes due to resorption. Resorption is most pronounced on the buccal side and might complicate implant placement as is could lead to proximity issues with the inferior alveolaris nerve of the mandible.

Alveolar ridge preservation (ARP) is commonly performed technique aimed at preserving available bone after tooth extraction. It facilitates delayed implant placement, reducing morbidity and providing optimal esthetic outcomes for implant placement. This procedure is performed using autogenous bone grafts, bone substitutes such as xenografts or allografts or a mixture of both. Also, membranes can be used to direct the growth of new bone.

A thin buccal bone wall is an indicator for bone loss that may compromise the integrity of the buccal bone and lead to biologic and esthetic complications. When the buccal bone wall has a width of < 1.5mm, it is considered an indication for ARP.

ARP is found to be effective in reducing bone loss and facilitating implant placement after extraction in the anterior region and for multi-rooted sides. However, most available evidence including RCTs, involves patients with at least 50% of buccal bone intact. Consequently, it is uncertain whether the efficacy ARP is also applicable in situations involving damaged sockets (buccal bone loss >50%).

ELIGIBILITY:
Inclusion Criteria:

* A minimum age of 18 years old
* In need for extraction of a single (pre)molar in the mandible that needs to be replaced by an implant
* At least one adjacent tooth
* A buccal bone defect after extraction of 50% or more

Exclusion Criteria:

* Active periodontal disease
* Uncontrolled diabetes mellitus
* History of or current chemotherapy or radiation in the head and neck area
* History of or current use of medication related to osteonecrosis of the jaw
* Heavy and moderate smokers (>5 cigarettes a day)
* Unable to maintain basic oral health (physical and/or mental)
* Pregnancy (in case of pregnancy, the treatment is postponed until after the delivery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2035-06-01 (Estimated); Study Completion 2035-06-01 (Estimated)

PRIMARY OUTCOMES:
The frequency of additional bone augmentation at implant placement. | During implant placement
  The frequency of additional bone augmentation at implant placement will be assessed during implant placement.

SECONDARY OUTCOMES:
Implant survival | From the moment of implant placement until 10 years of loading
  Implant survival is achieved if there is no presence of any mobility of the individual implant and/or any situation dictating implant removal.
Profilometric outcome measure | after intake, extraction, implant placement, placement of the final crown (after 2 weeks, 1 year, 3 years, 5 years and 10 years)
  Volumetric changes of the soft tissue
Prosthetic success | from placement of the final crown until 10 years of loading
  Prosthetic complications will be scored based on the modified United States Public Health Services (USPHS) criteria assessing framework fracture, veneering fracture, occlusal wear, marginal adaptation, anatomical form, cementation gap and patient satisfaction (Bayne & Schmalz, 2005). Suprastructures scoring delta will be scored as a failure. A suprastructure is scored as successful if all aspects scored only in the alpha or bravo categories (Pol et al., 2022).
Histological outcome measures | After implant placement
  Histological analysis
  Micro-computed tomography (μCT) analysis
Subjective Clinician-reported outcome measures related to the clinician's perception | After the surgical procedures (extraction and implant placement)
  Clinician questionnaire using an 11-point numeric scale assessing difficulty of the procedure. The lowest score is 0 which indicates extremely easy, the highest score is 10 which indicates extremely hard.
PROMS | at intake, after extraction, after implant placement, and 2 weeks, 1 year, 3 years, 5 years and 10 years after placement of the final crown
  Patient questionnaire based on a visual analog scales (VAS) score (0-10) assessing participant satisfaction evaluation during the study will be evaluated that will focus on satisfaction and impact of the surgical procedure and the aesthetic and functional result of the final crown. Score 0 indicates 'least agree' and score 10 indicates 'fully agree'.
Chair Time | At all surgical procedures (extraction, ARP, implant placement)
  Chair time in minutes
Costs | After 10 years of loading
  Costs in euros
Implant success | From one year after implant placement until 10 years of loading
  Absence of mobility, absence of persistent subjective complaints (pain, foreign body sensation and/or dysesthesia), absence of recurrent peri-implant infection with suppuration, absence of a continuous radiolucency around the implant, the annual vertical bone loss should not exceed 0.2 mm after the first year of service which should not exceed 1.5 mm, no pocket probing depth (PPD) of 5 mm or more with bleeding on probing (BOP) and no PPD of >5 mm.
Keratinized mucosal width (KMW) | 1-4 weeks, 1 year, 3 years, 5 years and 10 years after placement of the final crown.
  The width of the attached mucosa on the buccal side measured in the middle of the crown
Pocket probing depth (PPD) | 1-4 weeks, 1 year, 3 years, 5 years and 10 years after placement of the final crown
  The distance between the marginal gingival border and the tip of the pocket probe inserted against the implant (mesiobuccal, buccal, distobuccal, mesiopalatal, palatal, distopalatal)
Bleeding on probing (BOP) | 1-4 weeks, 1 year, 3 years, 5 years and 10 years after placement of the final crown
  Dichotomously (yes/no) at the mesiobuccal, buccal, distobuccal, mesiopalatal, palatal, distopalatal side of the implant.
Surgical complications (swelling, dehiscence, haemorrhage, infection) | 2 weeks post extraction and implant placement
  swelling (0= no visible oedema, 1 =slight oedema, 2= moderate oedema, 3= severe oedema), mucosal dehiscence (no dehiscence /small dehiscence of less than 2 mm/extensive dehiscence of more than 2mm) haemorrhage (absent/present) and infection (absent/present).
Marginal bone levels (MBL) | Post implant placement and 1, 3, 5 and 10 years after placement of the final crown.
  Changes in marginal bone level
Volumetric changes of the bone | after extraction, before implant placement, 1 year, 3 years, 5 years and 10 years after placement of the final crown
  Volumetric changes of the bone in percentage
Orofacial Esthetic Scale (OES-NL) | 2-4 weeks after placement, and 1, 3, 5 and 10 years after loading of the final crown
  Orofacial Esthetic Scale in Dutch(OES-NL) questionnaire assessing the esthetics of the teeth. Score 0 indicates very unsatisfied and score 10 indicates highly satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: J. Pijpe, Dr., MD, DDS, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avila-Ortiz G, Gubler M, Romero-Bustillos M, Nicholas CL, Zimmerman MB, Barwacz CA. Efficacy of Alveolar Ridge Preservation: A Randomized Controlled Trial. J Dent Res. 2020 Apr;99(4):402-409. doi: 10.1177/0022034520905660. Epub 2020 Feb 12. PMID 32050833
- [Background] Avila-Ortiz G, Chambrone L, Vignoletti F. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:195-223. doi: 10.1111/jcpe.13057. Erratum In: J Clin Periodontol. 2020 Jan;47(1):129. doi: 10.1111/jcpe.13212. PMID 30623987
- [Background] Monje A, Roccuzzo A, Buser D, Wang HL. Influence of buccal bone wall thickness on the peri-implant hard and soft tissue dimensional changes: A systematic review. Clin Oral Implants Res. 2023 Sep;34 Suppl 26:8-27. doi: 10.1111/clr.14177. PMID 37750522
- [Background] Pietrokovski J, Massler M. Alveolar ridge resorption following tooth extraction. J Prosthet Dent. 1967 Jan;17(1):21-7. doi: 10.1016/0022-3913(67)90046-7. No abstract available. PMID 5224784
- [Background] Van der Weijden F, Dell'Acqua F, Slot DE. Alveolar bone dimensional changes of post-extraction sockets in humans: a systematic review. J Clin Periodontol. 2009 Dec;36(12):1048-58. doi: 10.1111/j.1600-051X.2009.01482.x. PMID 19929956
- [Background] Jonker BP, Strauss FJ, Naenni N, Jung RE, Wolvius EB, Pijpe J. Early implant placement with or without alveolar ridge preservation in single tooth gaps renders similar esthetic, clinical and patient-reported outcome measures: One-year results of a randomized clinical trial. Clin Oral Implants Res. 2021 Sep;32(9):1041-1051. doi: 10.1111/clr.13796. Epub 2021 Jul 3. PMID 34129708
- [Background] Atieh MA, Alnaqbi M, Abdunabi F, Lin L, Alsabeeha NHM. Alveolar ridge preservation in extraction sockets of periodontally compromised teeth: A systematic review and meta-analysis. Clin Oral Implants Res. 2022 Sep;33(9):869-885. doi: 10.1111/clr.13975. Epub 2022 Jul 21. PMID 35818637
- [Background] Tonetti MS, Jung RE, Avila-Ortiz G, Blanco J, Cosyn J, Fickl S, Figuero E, Goldstein M, Graziani F, Madianos P, Molina A, Nart J, Salvi GE, Sanz-Martin I, Thoma D, Van Assche N, Vignoletti F. Management of the extraction socket and timing of implant placement: Consensus report and clinical recommendations of group 3 of the XV European Workshop in Periodontology. J Clin Periodontol. 2019 Jun;46 Suppl 21:183-194. doi: 10.1111/jcpe.13131. PMID 31215112